CLINICAL TRIAL: NCT03796507
Title: Early Post-surgical Temozolomide Therapy in Patients With High-Grade Gliomas Admitted to Acute Rehabilitation: A Feasibility Study
Brief Title: Early Temozolomide in Patients With High-Grade Gliomas in Rehabilitation
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Hiring freeze of research personnel due to COVID pandemic
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kevin Walter, Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSRB00003258
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Glioma of Brain
MeSH Terms: interventions — Temozolomide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Temozolomide Arm (Experimental): This study will only include one treatment group who will receive oral temozolomide at 75 mg per square meter of body surface area daily for 21 days before progressing to standard chemoradiation treatment.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — oral temozolomide at 75 mg per square meter of body surface area daily for 21 days

SUMMARY:
The purpose of this study is to investigate the feasibility of a possible treatment regimen that could be used to delay tumor progression in patients with glioblastoma. The study is being conducted in patients who qualify for inpatient rehabilitation, as this population is particularly vulnerable to delays in initiation of chemoradiation and further tumor growth in the period between surgical resection and the start of treatment.

DETAILED DESCRIPTION:
This is a pilot study to evaluate the feasibility and safety of early postsurgical temozolomide therapy prior to initiation of standard chemoradiation regimen in patients with glioblastoma who undergo inpatient rehabilitation. The study will be conducted with adult patients who qualify for inpatient rehabilitation following surgical resection of pathologically confirmed Grade IV glioma. Patients will begin a 21-day cycle of temozolomide starting 14 days after surgery at 75mg per square meter of body surface area daily to serve as bridge therapy. Patients will then progress to receive standard therapy following their rehabilitation stay. Patients will be assessed for their ability to complete the chemotherapy protocol without dose-limiting toxicity as well as complete inpatient rehabilitation successfully. Additionally, we will be assessing for tumor progression between the time of surgery and the time of treatment initiation.

If this study shows the expected results, the research team plans to proceed to a larger trial assessing the efficacy of early TMZ in patients with glioblastoma (GBM) who are admitted to acute inpatient rehabilitation compared to the current standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, aged 18+
* Newly diagnosed World Health Organization (WHO) Grade IV glioma, confirmed on pathology
* Karnofsky Performance Score ≥ 60
* Subject has undergone biopsy, subtotal resection, or gross total resection of tumor
* Subject has been evaluated by physical therapy and thought to be a candidate for acute rehabilitation
* Subject must be accepted for admission on 5-1200 unit at Strong Memorial Hospital
* Subject must be able to provide informed consent
* Subject must meet the following laboratory parameters:

  * Absolute neutrophil count > 1.5 x103/uL
  * Platelet count > 140 x103/uL
  * Alanine transaminase < 135 U/L
  * Aspartate transaminase < 120 U/L

Exclusion Criteria:

* Subject has received previous treatment for high-grade glioma
* Subject has other active malignancy
* Subject is currently pregnant or breastfeeding
* Subject is a women of childbearing potential who is not using a reliable method of contraception
* Subject has history of hypersensitivity to temozolomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
The number of patient who fail to complete temozolomide (TMZ) | 1 month
  The number of subjects who fail to complete early TMZ plus inpatient rehabilitation for any reason, including adverse events or progression or patient withdrawal

SECONDARY OUTCOMES:
Mean functional independence measure (FIM) score | 1 month
  FIM is comprised of 18 items, grouped into 2 subscales -motor and cognition. Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item therefore the better the health outcome. The total score for the FIM instrument (the sum of the motor and cognition subscale scores) will be a value between 18 and 126.
Response rate to TMZ | 1 month
  The response rate to early TMZ will be evaluated by comparing the MRI of the head before and after one course using the Response Assessment in Neuro-Oncology (RANO) criteria. The response rate will be reported with a (two-sided) 90% confidence interval. The RANO criteria consists of 5 elements: T1 Gadolinium enhancing disease, T2/FLAIR assessment, new lesions, use of corticosteroids and clinical status. Patients will be categorized as complete response, partial response, stable disease or progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Walter, MD, Principal Investigator — University of Rochester Medical Center, Dept. of Neurosurgery
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided